CLINICAL TRIAL: NCT02534519
Title: Applicability of Whole Genome Sequencing for Human Blood Group Genotyping and Genetic Definition of New Alleles as Exemplified on References and the Two MNSs-variants: U- and Stones(a)+
Brief Title: Whole Genome Sequencing for Blood Group Genotyping and Definition as Exemplified on U- and St(a)+.
Acronym: Blood Genome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Blood Donation Service Zurich, SRC (Other)
Responsible Party: Principal Investigator, Christoph Gassner, Priv. Doz. Mag. Dr. rer. nat. Christoph Gassner, Blood Donation Service Zurich, SRC
Other Study IDs: KEK-ZH-Nr. 2014-0408
Record Dates: First submitted 2015-08-10; First posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Genetic Blood Group (bg) Polymorphism in U Negativity and St(a) of MNSs
MeSH Terms: interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Case-Control
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Two times 10 mL EDTA-anticoagulated whole blood and genomic DNA resulting from this amount.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- people negative in bg MNSs antigen U: Blood group (bg) system MNSs. Individuals with phenotype "U-". Homo- and heterozygous individuals may be considered.
  Interventions: Other: Whole Genome Sequencing (WGS)
- people positive in bg MNSs antigen St(a): Blood group (bg) system MNSs. Individuals with phenotype "St(a)+". Homo- and heterozygous individuals may be considered.
  Interventions: Other: Whole Genome Sequencing (WGS)

INTERVENTIONS:
Other: Whole Genome Sequencing (WGS) — There will be no interventions needed other than blood sampling (20 mL blood) in the course of routine blood donation (450 mL blood) for 8 out of 10 individuals planned to be included as specimen, or reference samples in the study.

SUMMARY:
No health condition(s) are studied. Genetic background of blood groups is studied. U- and Stones(a)+ ("Caucasian type") are used as proof-of-principle samples. Disease associations of all blood group genes investigated are very rare, e.g. < 1 among 1'000 Swiss individuals (see table 1), and are not to be expected in the course of this study.

Genomic DNA of 2 U- samples were both provided as blinded reference material from New York and Vienna blood centres, respectively. Both donors are lost for follow up, and although there is no documented evidence for refusal of the respective donors to use their material in research projects, samples still lack informed consent.

DETAILED DESCRIPTION:
All 34 human blood group systems have at least two antithetical antigens and are of potential relevance during pregnancy and transfusion. Fortunately for every day routine practice, immunizations to foreign antigens are rare. Still, incompatibilities may occur in all blood group systems and will then require typing for the respective blood group antigens.

Blood genotyping evolved as the method of choice, in cases when typing reagents are commercially unavailable, or blood is inaccessible (foetus). In databases, most entries of blood group genes lack representative polymorphism (e.g. number of alleles). Moreover, many blood group antigens are insufficiently described in their intronic and inter-genetic sequences. This is true for results of unequal crossing-overs, gene-conversions and large insertions/deletions between highly homologous genes, especially within the blood group systems of Rhesus, e.g. RhD/RhCE and MN/Ss, respectively. Only Whole Genome Sequencing (WGS) allows for resolution of both problems: it delivers the whole blood group genome of an individual, and simultaneously recognizes new blood group alleles, or haplotypes. This request for ethical approval wants to test this assumption.

The antigenic determinants U- and Stones(a)+ of the blood group system MNSs still lack full genetic description and will serve as challenging examples for the description of new alleles (haplotypes) caused by large ins/del mutations of the two highly homologous genes GYPA and B. Genomic DNA of 2 U- samples were both provided as blinded reference material from New York and Vienna blood centres, respectively. Both donors are lost for follow up, and although there is no documented evidence for refusal of the respective donors to use their material in research projects, samples still lack informed consent. Additional reference samples (n max=4), and samples with suspected Stones(a)+ (n max=4) will be recruited from Zurich blood donors with informed consent, only.

ELIGIBILITY:
Inclusion Criteria:

* Existing biomaterial (gDNA), or
* Existing health related data for blood group U- (n max=2) and eligible for (venous) blood sampling of 20 mL, or
* Existing blood group pheno- and genotyping data indicating St(a)+ and eligible for (venous) blood sampling of 20 mL (n max=2), or
* Adequate blood group profile serving as reference (n max =4 & n max =4'000) and eligible for (venous) blood sampling of 20 mL.

Exclusion Criteria:

* Ineligible for venous blood sampling of approx. 20 mL.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Genomic DNA of 2 U- samples were both provided as blinded reference material from New York and Vienna blood centres, respectively. Both donors are lost for follow up, and although there is no documented evidence for refusal of the respective donors to use their material in research projects, samples still lack informed consent. Additional reference samples (n max=4), and samples with suspected Stones(a)+ (n max=4) will be recruited from Zurich blood donors with informed consent, only
Sampling Method: Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Whole Genome Sequencing for the definition of genetic background for blood group antigens U-, St(a)+ | 2 year period
  During a 2 year time-period, whole genome sequencing data generation and analysis will be used for the analysis and description of the genetic background for the blood group antigens U negativity, and for St(a).

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Gassner, PhD, Principal Investigator — Blutspende Zürich, Dienstleistungszentrum
Locations (1):
- Blutpende Zürich, Dienstleistungszentrum, Schlieren, Canton of Zurich, Switzerland